CLINICAL TRIAL: NCT07029399
Title: A Phase 1, First-in-Human, Open-Label Study to Evaluate the Safety, Tolerability, PK, and Preliminary Anti-tumor Activity of the Novel Oral Selective CDK2/CDK4 Dual Degrader NKT5097 in Adults With Advanced/Metastatic Solid Tumors
Brief Title: A Study With NKT5097 for Adults With Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NiKang Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKT5097-101
Record Dates: First submitted 2025-05-28; First posted 2025-06-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: HR+ Breast Cancer; Triple Negative Breast Cancer (TNBC); CCNE1 Amplified Advanced Solid Tumors; HR+ HER2- Breast Cancer; Ovarian Cancer; Endometrial Cancer; Uterine Carcinosarcoma
Keywords: CCNE1; cyclin E1; triple negative breast cancer; TNBC; estrogen receptor positive; HER2-; breast cancer; advanced solid tumors; post CDK4/6i; HER2 expression
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose Escalation (Experimental): Escalation of orally administered NKT5097
  Interventions: Drug: NKT5097 CDK2/CDK4 dual degrader
- Part 2 Food Effect (Experimental): Orally administered NKT5097 with and without meal
  Interventions: Drug: NKT5097 CDK2/CDK4 dual degrader
- Part 3 Expansion (Experimental): Expansion of dose levels based upon safety and PK following Part 1 escalation.
  Interventions: Drug: NKT5097 CDK2/CDK4 dual degrader

INTERVENTIONS:
Drug: NKT5097 CDK2/CDK4 dual degrader — NKT5097 will be distributed in tablet form and dosed daily or twice a day

SUMMARY:
The goal of this open-label dose escalation and expansion study is to evaluate the safety and tolerability of NKT5097 in adults with advanced/metastatic tumors (emphasis on breast cancer and solid tumors with CCNE1 amplification). Main questions to answer include:

* What is the recommended dose for expansion and/or Phase 2
* What medical issues/symptoms do participants experience when taking NKT5097

DETAILED DESCRIPTION:
This First-in-Human, Open-Label Study to Evaluate the Safety, Tolerability, PK, and Preliminary Anti-tumor Activity of NKT5097, a novel dual protein degrader of CDK2 and CDK4, is split into 3 Parts:

Part 1: Dose Escalation in selected advanced/metastatic non-CNS primary solid tumors will be enrolled based on a projected total of 5 dose levels

Part 2: Food Effect Analysis: Subjects with solid tumors (as noted in Part 1) will be enrolled (by backfilling selected dose cohorts) to evaluate the effect of dosing with food on NKT5097.

Part 3: Tumor-specific Expansion: Subjects may be enrolled (by backfilling selected dose cohorts) into each selected tumor-specific cohort. One or more of these cohorts may be opened at the discretion of the Sponsor in consultation with the DEC

In addition to the above, the study will explore pharmacokinetics, various pharmacodynamic biomarkers, gene mutations, and tumor responses such as PFS and DOR.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Advanced unresectable or metastatic solid tumor
* Refractory to or unable to tolerate existing therapies (Part 1 & 2 only)
* Measurable or evaluable disease (Part 1 & 2 only)
* Eighteen years of age or older
* ECOG status of 0 or 1
* Adequate organ function
* Patients with female reproductive organs must be surgically sterile, post- menopausal or willing to use effective contraception per protocol
* Patients who are capable of insemination must be willing to use highly effective contraception and to refrain from sperm donation during treatment and for 28 days after the last dose
* Able to swallow oral meds
* Willing to provide tumor tissue

Exclusion Criteria:

* Advanced solid tumor that is a candidate for curative treatment
* History of another malignancy except for the following: adequately treated local basal cell or squamous carcinoma of the skin, in situ cervical cancer, adequately treated papillary noninvasive bladder cancer, other adequately treated Stage I or Stage II cancers currently in complete remission
* Not recovered from the effects of prior anticancer therapy
* Clinically significant cardiovascular event, including myocardial infarction, arterial thromboembolism, or cerebrovascular thromboembolism, within 6 months
* Known active CNS metastases and/or carcinomatous meningitis
* Active interstitial lung disease requiring treatment
* History of uveitis, retinopathy, or other clinically significant retinal disease
* Major surgery within 30 days of administration of first dose
* Active uncontrolled infectious disease
* Significant liver disease (Child Pugh class B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities as Assessed by CTCAE | From enrollment through end of safety monitoring period of 28 days from first dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) as defined by CTCAE Version 5 | From enrollment through end of treatment up to 2 years
Maximum concentration Cmax after a single dose and multiple doses | Day 1 and Day 15 of Cycle 1 (Cycle 1 is 28 days)
Area under the concentration-time curve (AUC last) after a single dose and multiple doses from first dose through the last timepoint with quantifiable concentration (Tlast) | Day 1 and Day 15 of Cycle 1 ((Cycle 1 is 28 days)
Maximum concentration (Cmax) when dosed with and without food | Day 1 and Day 2 of Cycle 1 (Cycle 1 is 28 days)
Area under the concentration-time curve (AUC last) when dosed with and without food from dosing through the last timepoint with quantifiable concentration (Tlast) | Day 1 through Day 3 of Cycle 1 (Cycle 1 is 28 days)
Time to maximum plasma concentration (Tmax) after a single dose and multiple doses | Day 1 through Day 3 and Day 15 of Cycle 1 (Cycle 1 is 28 days)
Investigator-assessed ORR by RECIST v1.1 | From enrollment (Day 1) through end of treatment (up to 3 years) with an average of 4 months
Investigator-assessed PFS by RECIST v1.1 | From enrollment (Day 1) through end of treatment (up to 3 years) with an average of 4 months
Duration of Response (DOR) | From enrollment (Day 1) through end of treatment (up to 3 years) with an average of 4 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - SCRI Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START) San Antonio, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics (START) Mountain Region, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No